CLINICAL TRIAL: NCT05111808
Title: A Non-Randomized, Prospective, Open Label, Single-site Feasibility Trial for Real-time Identification of the Ureters With a Methylene-blue fluoroPhore
Brief Title: Feasibility Trial for Real-time Identification of the Ureters With a Methylene-blue
Acronym: TRIUMPh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 120726
Record Dates: First submitted 2021-10-12; First posted 2021-11-08 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Fluorescence Guided Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methyl Blue (Experimental): This group will receive intraoperative IV methyl blue
  Interventions: Device: Methylene blue fluorescence

INTERVENTIONS:
Device: Methylene blue fluorescence — IV administration of methylene blue, detection with deep infrared camera and light source

SUMMARY:
This is a non-randomized prospective, open label, single site study to evaluate the feasibility of recruitment for the use of an Investigational Endoscopic Fluorescence Imaging System, PINPOINT, in intraoperative bilateral visualization of ureters using intravenous injection of methylene blue. Feasibility of urine sample collection during surgery will also be assessed.

DETAILED DESCRIPTION:
Background - During certain abdominal surgeries there is difficulty in finding the ureters, which act as a conduit for urine from the kidneys to the bladder. If the ureters are sectioned during surgery this causes great suffering for the patient and increased costs for the hospital and the National Health Service. Even experienced surgeons are at risk of causing this dreaded complication.

Methylene blue can emit a fluorescent signal and highlight the ureters in real time during surgical procedures. A study is necessary to evaluate the effectiveness of methylene blue fluorescence to identify the ureters during surgery.

Methods - In this study, patients undergoing abdominal surgery with high risk for ureter complications will be included. The feasibility of recruitment of these patients will be assessed using a screening log. Included patients with receive intraoperative methylene blue injection in increasing doses. Urine samples will be taken to establish the conversion of methylene blue to leucomethylene blue.

Expected results - the investigators expect to define the recruitment rate of the patient group of interest and to identify the causes for non recruitment. Secondary outcomes are ureteric identification and conversion of methylene blue to leucomethylene blue.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Scheduled for a surgery where routine ureter identification is used
* Have signed an approved informed consent form for the study
* Be willing and able to comply with the study protocol

Exclusion Criteria:

* Known allergy or history of adverse reaction to methylene blue
* Taking an antidepressant including, but not limited, to selective and non-selective serotonin reuptake inhibitors, or a psychiatric medication
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Renal dysfunction defined as estimated glomerular filtration rate (eGFR) of <60 mL/min/1.73 m2
* Has participated in another investigational study within 30 days prior to surgery
* Pregnant or lactating subjects
* Subjects who, in the Investigator's and/or designee's opinion, have any medical condition that makes the subject a poor candidate for the investigational procedure, or interferes with the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment to study | 12 months
  Feasibility of recruitment to the study. This will be recorded in the screening log. The number of patients able partake in the study will be expressed as a percentage of the number of patients approached for consent.
  Patients will be excluded if the do not meet the inclusion/exclusion criteria or do not consent.

SECONDARY OUTCOMES:
Rate of ureteric identification and signal intensity at defined time points | 12 months
  The operation will be paused and image switched to the Pinpoint camera at 5, 10, 15, 20, 30 and 40 minutes. The signal to background ratio will be calculated from the near infra-red images. This will allow us to quantify the fluorescence of methylene blue under near infra-red light.
Percentage conversion of methylene blue to leucomethylene blue at defined time points | 12 months
  Urine samples will be taken at 10 minute intervals after the administration of methyl blue. The ratio of methylene blue to leucomethylene blue will be calculated at each of these stages to determine the likely rate of conversion rate.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Chand, PhD, Principal Investigator — University College, London
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No